CLINICAL TRIAL: NCT04649021
Title: Safety and Immunogenicity of SARS-CoV-2 mRNA Vaccine (BNT162b2) in Chinese Healthy Population: A Phase II, Randomized, Placebo-controlled, Observer-blinded Study
Brief Title: Safety and Immunogenicity of SARS-CoV-2 mRNA Vaccine (BNT162b2) in Chinese Healthy Population
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Collaborators: Shanghai Fosun Pharmaceutical Industrial Development Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BNT162-06
Record Dates: First submitted 2020-11-17; First posted 2020-12-02 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: SARS-CoV-2
Keywords: Coronavirus Disease 2019; Coronavirus infection; Vaccine; Protection against COVID-19; Covid19; SARS (Severe Acute Respiratory Syndrome)
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Severe Acute Respiratory Syndrome | interventions — BNT162 Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BNT162b2 18-85 years of age (Experimental)
  Interventions: Biological: BNT162b2
- Placebo 18-85 years of age (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: BNT162b2 — Intramuscular injection
  Arms: BNT162b2 18-85 years of age
Other: Placebo — Intramuscular injection
  Arms: Placebo 18-85 years of age

SUMMARY:
This is a phase II, randomized, placebo-controlled, observer-blinded study of the safety and immunogenicity of SARS-CoV-2 messenger RNA (mRNA) vaccine (BNT162b2) in Chinese healthy population. After randomization, the trial for each participant will last for approximately 13 months. Screening period is 2 weeks prior to randomization (Day -14 to Day 0), and two doses of either SARS-CoV-2 vaccine (BNT162b2) or placebo will be given intramuscularly (IM) separated by 21 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants between the ages of 18 and 85 years, inclusive, at randomization.
* Participants who are willing and able to comply with all scheduled visits, vaccination plan, laboratory tests, lifestyle considerations, and other study procedures.
* Healthy participants who are determined by medical history, physical examination (if required), and clinical judgment of the investigator to be eligible for inclusion in the study. Note: Healthy participants with preexisting stable disease, defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 6 weeks before enrollment, can be included.
* Capable of giving personal signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form and this protocol.
* SARS-CoV-2 antibody test screening is negative.
* Negative SARS-CoV-2 test in throat swabs by reverse transcription-polymerase chain reaction (RT-PCR) (only for the first approximately 150 subjects).
* Normal in chest computed tomography (CT) scans (no imaging features of coronavirus disease 2019 (COVID-19), only for the first approximately 150 subjects).

Exclusion Criteria:

* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Known infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B virus (HBV).
* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention(s).
* Receipt of medications intended to prevent COVID-19.
* Immunocompromised individuals with known or suspected immunodeficiency, determined by history and/or laboratory/physical examination.
* Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
* Women who are pregnant or breastfeeding.
* Previous vaccination with any coronavirus vaccine.
* Individuals who receive treatment with immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids, eg, for cancer or an autoimmune disease, or planned receipt throughout the study. If systemic corticosteroids have been administered short term (<14 days) for treatment of an acute illness, participants should not be enrolled into the study until corticosteroid therapy has been discontinued for at least 28 days before study intervention administration. Inhaled/nebulized, intra-articular, intrabursal, or topical (skin or eyes) corticosteroids are permitted.
* Receipt of blood/plasma products or immunoglobulin, from 60 days before study intervention administration or planned receipt throughout the study.
* Participation in other studies involving study intervention within 28 days prior to study entry and/or during study participation.
* Previous participation in other studies involving study intervention containing lipid nanoparticles.
* Have had contact with confirmed COVID-19 patients or persons tested positive for SARS-CoV-2 within the 30 days prior to Screening Visit.
* Travel or live in any country or region with a high SARS-CoV-2 infection risk (as defined at Screening Visit) within the 14 days prior to Screening Visit.
* Symptoms of COVID-19, e.g., respiratory symptoms, fever, cough, shortness of breath and breathing difficulties.
* Fever, defined as axillary temperature ≥37.3ºC or oral temperature ≥38ºC.
* History of SARS, SARS-CoV-2 or middle east respiratory syndrome (MERS) infection. Suspected SARS patients should be screened for SARS antibodies.
* Investigator site staff or Fosun employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 950 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2021-02-07 (Actual); Study Completion 2022-01-09 (Actual)

PRIMARY OUTCOMES:
SARS-CoV-2 serum neutralizing titers - Seroconversion rates (SCR) | 1 Month after Dose 2
  SCR of SARS-CoV-2 serum neutralizing titers at 1-month after dose 2. Seroconversion is defined as ≥4-fold rise from before vaccination to 1-month post dose 2.
The geometric mean titer (GMT) of SARS-CoV-2 serum neutralizing titers at 1 month after dose 2 | 1 Month after Dose 2

SECONDARY OUTCOMES:
SARS-CoV-2 serum neutralizing titers - SCR | 1 Week, 6 and 12 Months after Dose 2
  Compared with baseline before Vaccination 1, SCR of SARS-CoV-2 serum neutralizing titers at 1 week, 6 and 12 months after dose 2.
SARS-CoV-2 serum neutralizing titers - GMT | 1 Week, 6 and 12 Months after Dose 2
  GMT of SARS-CoV-2 serum neutralizing titers at 1 week, 6 and 12 months after dose 2.
SARS-CoV-2 anti-S1 immunoglobulin G (IgG) antibody level - SCR | 1 Week, 1, 6 and 12 Months after Dose 2
  Compared with baseline before Vaccination 1, SCR of SARS-CoV-2 anti-S1 IgG antibody level at 1 week, 1, 6 and 12 months after dose 2.
SARS-CoV-2 anti-S1 IgG antibody level - GMT | 1 Week, 1, 6 and 12 Months after Dose 2
  GMT of SARS-CoV-2 anti-S1 IgG antibody level at 1 week, 1, 6 and 12 months after dose 2.
SARS-CoV-2 serum neutralizing antibody level - Geometric mean fold rise (GMFR) | 1 Week, 1, 6 and 12 Months after Dose 2
  Compared with baseline before Vaccination 1, the GMFR of SARS-CoV-2 serum neutralizing antibody titers at 1 week, 1, 6 and 12 months after dose 2.
SARS-CoV-2 anti-S1 IgG antibody level - GMFR | 1 Week, 1, 6 and 12 Months after Dose 2
  Compared with baseline before Vaccination 1, GMFR of SARS-CoV-2 anti-S1 IgG antibody level at 1 week, 1, 6 and 12 months after dose 2.
Percentage of participants reporting local reactions | Within 7 Days and 14 Days after each vaccination
  Pain at the injection site, redness, and swelling as self-reported on diary cards.
Percentage of participants reporting systemic events | Within 7 Days and 14 Days after each vaccination
  Fever, fatigue, headache, chills, vomiting, diarrhea, new or worsened muscle pain, and new or worsened joint pain as self-reported on diary cards.
Hematology laboratory assessments | Day 1 and 7 Days after Dose 1, before Dose 2, and 7 Days after Dose 2
  Percentage of participants with abnormal hematology laboratory values 1 and 7 days after dose 1, before dose 2, and 7 days after dose 2.
Chemistry laboratory assessments | Day 1 and 7 Days after Dose 1, before Dose 2, and 7 Days after Dose 2
  Percentage of participants with abnormal chemistry laboratory values 1 and 7 days after dose 1, before dose 2, and 7 days after dose 2.
Hematology laboratory assessments | Day 1 and 7 Days after Dose 1; and before Dose 2 and 7 Days after Dose 2
  Percentage of participants with grading shifts in hematology laboratory assessments between baseline and 1 and 7 days after dose 1; and before dose 2 and 7 days after dose 2.
Chemistry laboratory assessments | Day 1 and 7 Days after Dose 1; and before Dose 2 and 7 Days after Dose 2
  Percentage of participants with grading shifts in chemistry laboratory assessments between baseline and 1 and 7 days after dose 1; and before dose 2 and 7 days after dose 2.
Adverse events (AEs) | From Dose 1 through 1 Month after the last Dose
  AEs from dose 1 to 1 month after the last dose.
Serious AEs (SAEs) | From Dose 1 through 6 Months after the last Dose
  SAEs from dose 1 to 6 months after the last dose.

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (1):
- Jiangsu Provincial Center for Disease Control and Prevention, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hui AM, Li J, Zhu L, Tang R, Ye H, Lin M, Ge L, Wang X, Peng F, Wu Z, Guo X, Shi Y, Pan H, Zhu J, Song Z, Qiu J, Wang W, Zheng J, Ozhelvaci O, Shpyro S, Bushway M, Derhovanessian E, Kuhnle MC, Luxemburger U, Muik A, Shishkova Y, Khondker Z, Hu S, Lagkadinou E, Sahin U, Tureci O, Zhu F. Immunogenicity and safety of BNT162b2 mRNA vaccine in Chinese adults: A phase 2 randomised clinical trial. Lancet Reg Health West Pac. 2022 Dec;29:100586. doi: 10.1016/j.lanwpc.2022.100586. Epub 2022 Sep 14. PMID 36120090